CLINICAL TRIAL: NCT02845635
Title: MS Mosaic: A Longitudinal Research Study on Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00072319
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Relapsing Remitting Multiple Sclerosis: Those who document during the study on-boarding process that they suffer from relapsing-remitting multiple sclerosis.
  Interventions: Other: Personal history of multiple sclerosis
- Primary Progressive Multiple Sclerosis: This who document during the on-boarding process that they suffer from primary progressive multiple sclerosis.
  Interventions: Other: Personal history of multiple sclerosis
- Secondary Progressive Multiple Sclerosis: This who document during the on-boarding process that they suffer from secondary progressive multiple sclerosis.
  Interventions: Other: Personal history of multiple sclerosis
- Control: This who document during the on-boarding process that they do not suffer from multiple sclerosis.
  Interventions: Other: Personal history of multiple sclerosis

INTERVENTIONS:
Other: Personal history of multiple sclerosis — Participants will be stratified into one of four cohorts based on their experience (or lack of experience) with the three major forms of multiple sclerosis.

SUMMARY:
The purpose of this study is to better characterize the fluctuations in multiple sclerosis symptoms and their relationship to medications, to length/extent of disease, and to a variety of physiologic measures.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Live in the United States of America
* Read/write in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be self-selecting from the national release of a mobile application.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change in perceived fatigue severity (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in perceived cognitive impairment (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
  Severity of cognitive impairment experienced from multiple sclerosis
Change in perceived depression or anxiety severity (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
  Severity of any mood disorders experienced from multiple sclerosis

SECONDARY OUTCOMES:
Change in perceived walking instability (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in perceived vision difficulties (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in perceived Bowel/Bladder dysfunction (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
  Severity of bowel/bladder dysfunction experienced from multiple sclerosis
Change in perceived sensory disturbance (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in perceived vertigo severity (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in perceived dysarthria severity (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in pain (self-report) as recorded by symptom diary | Every 24 hours through study completion, an average of 6 months
Change in sleep quality as recorded by app-linked wearable device | Every 24 hours through study completion, an average of 6 months
Change in medication adherence (self-report) as recorded by medication diary | Every 24 hours through study completion, an average of 6 months
Change in self-efficacy (self-report) as determined by the Multiple Sclerosis self-efficacy scale (survey instrument) | every three months, through study completion (an average of 6 months)
Change in Multiple Sclerosis Quality of Life Inventory | prompted based on the app user's responses on the daily surveys, up to 6 months
  The Multiple Sclerosis Quality of Life Inventory surveys are prompted based on the app user's responses on the daily surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Fletcher L Hartsell, MD MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No